CLINICAL TRIAL: NCT03556930
Title: Simulated Radiotherapy Treatment Assisted With Pediatric Radiation Oncology With Movie Induced Sedation Effect (PROMISE) Technique
Brief Title: Simulated Radiotherapy Treatment Assisted With Pediatric Radiation Oncology With Movie Induced Sedation Effect Technique
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Project was never initiated.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU 042018-088
Record Dates: First submitted 2018-05-18; First posted 2018-06-14 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Childhood Cancer
Keywords: Non-sedated radiotherapy treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Movie Induced Sedation Effect (Experimental): Pediatric Radiation Oncology with Movie Induced Sedation Effect monitored by an AlignRT system (VisionRT LTD, UK).
  Interventions: Device: AlignRT system (VisionRT LTD, UK)

INTERVENTIONS:
Device: AlignRT system (VisionRT LTD, UK) — Pediatric patient will watch age-proper movie during radiation treatment. The motion of pediatric patient will continually be monitored by an AlignRT system (VisionRT LTD, UK). Both movie and radiation beam will be paused if the motion of pediatric patient is beyond positioning accuracy threshold. Movie and beam will be resumed if pediatric patient is positioning with in tolerance.

SUMMARY:
Pediatric patient will watch age-proper movie during radiation treatment. The motion of pedi-patient will continually be monitored by an AlignRT system (VisionRT LTD, UK).

DETAILED DESCRIPTION:
For most pediatric cancer patients under 7 years of age, current standard radiotherapy practice involves the use of anesthesia or sedation at each fraction to ensure that the patient remains still during the treatment. A child may receive up to 30 episodes of anesthesia in succession. This also means that, for the 6-week duration of radiotherapy, a child may never fully return to his/her baseline activity. More importantly, the excessive use of anesthesia introduces many risks and side effects that, combined with chemotherapy, and cancer itself, can greatly reduce the overall treatment experience for the children and their families

In the two years, the investigators have been actively developing technologies to facilitate a novel pediatric radiotherapy, which called Pediatric Radiation Oncology with Movie Induced Sedation Effect (PROMISE). The main idea of PROMISE is that pediatric patient will watch age-proper movie during radiation treatment. The motion of pediatric patient will continually be monitored by an AlignRT system (VisionRT LTD, UK). Both movie and radiation beam will be paused if the motion of pediatric patient is beyond positioning accuracy threshold. Movie and beam will be resumed if pediatric patient is positioning with in tolerance.

In this study, the investigators will use the developed PROMISE software and hardware platform to evaluate the feasibility of non-sedated radiotherapy treatment.

The investigator will use radio to mimic radiation beam delivery and gantry motion to mimic radiation device rotation. Pediatric patient will watch an age-appropriate movie of his/her choice. AlignRT (VisionRT LTD, UK) imaging system will be used to monitor the motion of the patient. If the motion exceeds any pre-defined positioning thresholds the sound mimic treatment beam noise will be held off and the movie will be paused.

If the patient reverts to treatment position within a pre-defined temporal threshold (1 minute), the simulated treatment will be resumed with a continuing movie.

If the patient cannot revert to the treatment position within a pre-defined time threshold/or the movement is beyond any pre-defined re-alignment threshold value the radiation beam and the movie will be turned off, the patient will be readjusted and the treatment will resume.

In any study case, the simulated PROMISE treatment will be ceased if therapists have to re-position the patient more than three times.

The simulated PROMISE treatment will be repeated in three times in three different days.

ELIGIBILITY:
Inclusion Criteria:

Patients Age: ≥4 and ≤10

Patients and his/her legal guardian must be willing and capable to provide informed consent to participate in the protocol.

Patients must be compliant to all required pretreatment evaluations:

1. Informed Consent
2. Medical Diagnosis
3. Demographics
4. Review subject eligibility criteria
5. Physical exam including vital signs, height and weight Vital signs (temperature, pulse, respirations, blood pressure) will be collected before simulation treatment.
6. Simulated PROMISE treatment screening Patient will be asked for lying on treatment couch for 30 seconds with PROMISE movie on. If patient stay still for 30 seconds, s/he is eligible for the simulated PROMISE treatment

Exclusion Criteria:

Patients aren't compliant to all required pretreatment evaluations

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
To investigate the feasibility of applying PROMISE for pediatric radiotherapy by analyzing overall treatment time | in three different days
  Analyze overall treatment time including time for hardware and software setup

SECONDARY OUTCOMES:
To determine overall PROMISE radiotherapy treatment efficiency | in three different days
  - Analyze PROMISE workflow based on record time:
  Times of beam/movie pauses. Times the child reverts back to the treatment position.
To quantify PROMISE radiotherapy treatment dose deviation | in three different days
  - Analyze the dose deviation from original treatment plan.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Jiang, Ph.D, Principal Investigator — University of Texas Southwestern Medical Center